CLINICAL TRIAL: NCT01378026
Title: Study of the Role of G72 in Amyotrophic Lateral Sclerosis: Biomarker Discovery and Mechanism Investigation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Hao-Teng Chang, Ph.D., China Medical University
Other Study IDs: DMR100-IRB-069
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Amyotrophic Lateral Sclerosis; Alzheimer Disease; Parkinson's Disease
Keywords: Amyotrophic Lateral Sclerosis; G72; SNP
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood, serum and DNA

SUMMARY:
G72 gene is located on the common linkage locus in bipolar disorder and schizophrenia, and it encodes D-amino acid oxidase activator (DAOA). There are evidences that elucidated G72 and D-amino acid oxidase(DAO) together playing a critical role in the pathophysiology of schizophrenia. Recently, reports discovered missense mutations in the DAO (R199W DAO and R38H DAO) are associated with familial amyotrophic lateral sclerosis (FALS), and our preliminary data showed that the level of G72 autoantibody decreases in patients with ALS compared with normal control. Thus, we want to find out whether G72 plays a role in ALS and neurodegenerative diseases including Alzheimer disease and Parkinson's disease. First, we detect G72 protein and its autoantibody in sera of neurodegenerative diseases patients using ELISA and Western blotting, and the data are compared with normal control. We hypothesize the levels of G72 protein and its autoantibody in neurodegenerative diseases are less than those in normal control. Then, we extract genomic DNA of neurodegenerative diseases patients, and use polymerase chain reaction(PCR) to detect single nucleotide polymorphism (SNP) of G72. We aim to detect G72 missense SNP variants presented in ALS, AD and PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease, Parkinson's disease and amyotrophic lateral sclerosis

Exclusion Criteria:

-

Ages: 32 Years to 87 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients were from Taipei city hospital-ZhongXiao branch.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-01